CLINICAL TRIAL: NCT04719260
Title: Nutrition Thinking® Randomized Clinical Trial for Scientific Validation of a Nutritional Approach Based on the Values and Methodology of Design Thinking
Brief Title: Nutrition Thinking® Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Mauricio Kunz (Unknown); Caroline Nespolo de David (Unknown); Renato Gorga Bandeira de Mello (Unknown); Aline Marcadenti de Oliveira (Unknown)
Responsible Party: Principal Investigator, Francisca Mosele, Principal Investigator, Hospital de Clinicas de Porto Alegre
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-0694
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Overweight
Keywords: nutrition thinking; nutritional approach; diet; design thinking; overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: This is a parallel randomized clinical trial, where individuals will be allocated to one of the arms - experimental intervention (Nutrition Thinking®) or control (standard intervention) - in a 1:1 ratio. The sample size calculation suggests that 82 subjects (41/each arm) are required. At the end of the clinical trial, individuals will be part of a cohort study where they will be followed up every three months for 12 months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be generated by computer in the data center using alphanumeric codes and implemented through the Research Electronic Data Capture (REDCap®) software. The professionals who will carry out the interventions during the protocol will be trained for one of the two interventions, without knowledge of the outcomes (except, bioimpedance results), evaluations performed during the study or comparison intervention. After the assignment to one of the groups, the participants, and those who will evaluate all the outcomes, will remain blind until the end of the study and results analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition Thinking® (Experimental): Nutrition Thinking® approach to promote weight loss and healthy diet pattern.
  Interventions: Behavioral: Nutrition Thinking®
- Standard Nutritional Approach (Active Comparator): The traditional nutritional prescriptive approach.
  Interventions: Behavioral: Standard Nutritional Approach

INTERVENTIONS:
Behavioral: Nutrition Thinking® — In the first session, the nutritionist will carry out the anamnesis through the Empathy Map and assessment of the nutritional status to define the Nutrition Briefing. The steps described by Design Thinking as understanding, observation, and point of view comprise the first phase of this session. The ideation process will proceed from the definition of the Nutrition Challenge. Prototyping is the final stage of the first session, where an initial prototype of the diet will be co-created based on visual thinking tools and the description underlying the creation of diets. Within 24 hours the individual will receive a summary of the material developed by email. The period between sessions will comprise the testing phase and the follow-up sessions the iteration phase where the experience and previous steps are revisited in order to create new insights, anthropometric measurements will be seen as reflections of the experience and not as primary outcomes of the intervention.
  Arms: Nutrition Thinking®
Behavioral: Standard Nutritional Approach — In the first session the nutritionist will carry out the food and nutritional anamnesis and assessment of the nutritional status. From this information, the nutritionist will generate the diagnostic hypothesis and determine the specific nutritional needs. The professional will be responsible for generating the dietary prescription defining the characteristics of the diet that will be delivered printed to the individual after a period of 15 days, in the second session of the protocol. The follow-up session will be based on adherence to the established conduct and monitoring of anthropometric variations.
  Arms: Standard Nutritional Approach

SUMMARY:
The purpose of this study is to scientifically validate Nutrition Thinking®, a novel nutritional approach based on the values and methodologies of Design Thinking.

DETAILED DESCRIPTION:
The concept of nutrition has changed exponentially in recent decades to include a range of challenges that were not foreseen. The strength of this movement is based on the understanding of (1) the complexity with which people face their nutritional challenges; and (2) the interconnection between food systems and overlapping health risks associated with malnutrition, obesity, and climate change.

Maintaining an adequate weight, a healthy and sustainable diet pattern are complex well-established challenges. However, current nutritional approaches to lose weight, based on functional experiences, often fail to promote long-term adherence to dietary recommendations and maintaining lost weight.

The ambiguity and complexity that involves an interactional nutrition, based on the experiences involved in how people act at the individual level and their relationships with the environment and dynamic systems, brings up the challenge of designing meaningful learning experiences to promote a change of culture and positive impact.

Current social changes demand the search for novel nutritional approaches based on methodologies that result in meaningful experiences. We need new ways to build diets that balance the needs of individuals and society as a whole, new ideas that address global challenges, new strategies that result in differences that matter, and a sense of purpose that includes everyone involved.

With that in mind, Nutrition Thinking® arises as a nutritional approach based on the values and methodologies of Design Thinking, an abstraction of a mental model for addressing complex problems and conducting projects based on empathy, collaboration, and experimentation. Therefore, Nutrition Thinking® represents a new nutrition learning matrix based on experience for the co-creation of authentic and sustainable diets.

ELIGIBILITY:
Inclusion Criteria:

* age between 25 and 35 years old of both sexes;
* nutritional diagnosis of overweight (BMI between 25-29.9 kg/m2);
* available to participate in the sessions proposed by the protocol (every 15 days for a period of 3 months).

Exclusion Criteria:

* presence of characteristics that make nutritional assessment impossible (eg. presence of metallic prostheses or amputated limbs);
* previous involvement in any clinical trial, nutritional or medical intervention for weight loss in the 6 months prior to recruitment;
* previous history of eating disorders (anorexia, bulimia, binge eating);
* presence of congenital diseases;
* presence of thyroid disease, hypertension, dyslipidemia and diabetes, defined through medical diagnosis associated with drug treatment and / or previous or current cardiovascular disease;
* pregnant or lactating women.

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks
  Weight change from baseline to end of intervention
Quality of diet | 12 weeks
  Changes in The Healthy Eating Index 2015 score (HEI-2015) from baseline to end of intervention. The Healthy Eating Index-2015 (HEI-2015) allows us to assess how well a set of foods aligns with the 2015-2020 Dietary Guidelines for Americans. The HEI-2015 includes 13 components that can be summed to a maximum total score of 100 points. The components capture adequacy components and moderation components. For the adequacy components, higher scores reflect higher intakes that meet or exceed the standards. For the moderation components, higher scores reflect lower intakes because lower intakes are more desirable. A higher total score indicates a diet that aligns better with the Dietary Guidelines. Adequacy components include total fruits, whole fruits, total vegetables, greens and beans, whole grains, dairy, total protein foods, seafood and plant proteins, fatty acids. Moderation components include refined grains, sodium, added sugars, and saturated fats.
Dietary usability | 12 weeks
  Dietary usability will be measured by the System Usability Scale (SUS). The SUS consists of ten statements. For each statement, the participant gives his or her approval or rejection in the form of a scale ranging from 1=strong approval to 5=strong rejection of the statement. The results of the SUS questionnaire are used to calculate a numerical value (the so-called SUS score). The categories in the SUS questionnaire are coded with values from 0 to 4. The results can have a value between 0 (worst application imaginable) and 100 (best application imaginable): when the questionnaire is evaluated, the numbers obtained are added together - the sum is between 0 and 40 - and then multiplied by 2.5 and will be normalized to produce a percentile ranking.

SECONDARY OUTCOMES:
Food literacy | 12 weeks
  Food literacy changes from baseline to end of intervention will be defined by the Short Food Literacy Questionnaire (SQLF). The SQLF employed a Likert-type scale to measure individual item scores and summed to create a composite score minimum score 7 points, maximum 52 points. Higher scores are associated with a better level of literacy in food.
Body fat percentage | 12 weeks
  Body fat percentage change from baseline to end of intervention will be measured with multi-frequency segmental bioelectrical impedance.
Carbon Footprint | 12 weeks
  Carbon footprint (CF) change from baseline to end of intervention will be estimated through individual-level carbon footprints (ICF) are assessed as ICF = ΣCiEi where each term is the product of the degree of consumption © and the CO2 equivalent radiative forcing emission (E) of that input (i). Greenhouse gas emission (E) weightings applied to individual consumption levels (C) will be expressed in metric tons CO2-equivalent/year (CO2e).

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Mosele, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Muricio Kunz, PhD, Study Chair — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No